CLINICAL TRIAL: NCT07383363
Title: Comparison of Efficacy and Safety of Vita 6 Versus Zinc Along With Applied Behavioural Therapy in Management of Autism Spectrum Disorder in Children Aged 3-14 Years
Brief Title: Comparison of Efficacy and Safety of Vita 6 Versus Zinc Along With Applied Behavioural Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Nadeem-Multan
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vita 6 Group (Experimental): Patients will be given one tablet of Vita 6 (50 mg) twice a day for 3 months, along with applied behavioral therapy.
  Interventions: Drug: Vita 6
- Zinc Group (Experimental): Patients will receive syrup zinc sulfate 2 mg/kg/day as a single dose for 3 months, along with applied behavioral therapy.
  Interventions: Drug: Zinc sulfate

INTERVENTIONS:
Drug: Vita 6 — Patients will be given one tablet of Vita 6 (50 mg) twice a day for 3 months, along with applied behavioral therapy.
  Arms: Vita 6 Group
Drug: Zinc sulfate — Patients will receive syrup zinc sulfate 2 mg/kg/day as a single dose for 3 months, along with applied behavioral therapy.
  Arms: Zinc Group

SUMMARY:
The study seeks to fill the gaps in available local data regarding the diagnosis and its management, as multiple treatments are in practice. Therefore, the study aimed at the comparison of efficacy and safety of Vita 6 versus zinc along with applied behavioral therapy in the management of autism spectrum disorder in children aged 3-14 years.

DETAILED DESCRIPTION:
Although autism spectrum disorder is a genetic disorder, environmental factors can play a role in its etiology. Local people and doctors now know about autism but have less knowledge about how to diagnose it and its management. Although its mainstay of treatment is applied behavioral therapy, a few medicines like Vita 6, zinc folinic acid, and methylcobalamin are now under trial in its management with favorable results. Since literature shows variable treatment outcomes for these medications, the findings would help clinicians to opt for a medication capable of reducing the severity of the symptoms with safety and economy.

ELIGIBILITY:
Inclusion Criteria:

* Children of any gender
* Aged 3-12 years
* Newly diagnosed patients of autism spectrum disorder following the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria
* Not taking any treatment

Exclusion Criteria:

* With any of psychiatric disorder
* With any of movement disorder

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
Reduction in severity | 3 months
  Efficacy of the treatment will be assessed using the Childhood Autism Rating Scale (CARS) score, which ranges between 15 and 60. Efficacy will be deemed 'yes' if a CARS score lower than the baseline is achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Iqbal, Principal Investigator — Children's Hospital and institute of Child Health Multan, Punjab, Pakistan; Erum Afzal, FCPS, Study Director — Children's Hospital and institute of Child Health Multan, Punjab, Pakistan
Locations (1):
- Children Hospital and Institute of Child Health, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.